CLINICAL TRIAL: NCT01131325
Title: A Multi-center, Single Arm Study of Nilotinib in Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP) Patients With Low Imatinib Trough Plasma Concentrations
Brief Title: Study of Nilotinib in Ph+ CML-CP Patients With Low Imatinib Trough Plasma Concentrations
Acronym: MACS1148
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107AUS20
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Results first posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2020-10

CONDITIONS: CML; Philadelphia Chromosome Positive (Ph+); Chronic Myelogenous Leukemia Chronic Phase(CML-CP) Patients With Low Imatinib Trough Levels
Keywords: Philadelphia chromosome positive; Ph+; chronic myelogenous leukemia chronic phase; CML-CP; low imatinib trough levels
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nilotinib (Experimental)
  Interventions: Drug: nilotinib

INTERVENTIONS:
Drug: nilotinib — All patients will receive nilotinib 300mg bid po daily. Nilotinib dose is taken every 12 hours
  Other Names: AMN107; Tasigna

SUMMARY:
This study is to determine the number of European Leukemia Network (ELN)guideline defined treatment failure events from time of study entry in CML-CP patients with low imatinib trough concentrations treated with nilotinib.

ELIGIBILITY:
Inclusion Criteria:

* Cytogenetically confirmed Ph+ CML-CP Any prior dose of Imatinib
* Imatinib 400 mg daily for ≥7 consecutive days prior to imatinib trough collection
* Imatinib trough plasma concentration <850 ng/mL

Exclusion Criteria:

* Prior documented failure events as defined by ELN guidelines:
* Loss of CHR, CCyR, or clonal progression/Ph+
* Less than CHR at 3 months after diagnosis
* No CyR at 6 months after diagnosis
* Less than PCyR at 12 months after diagnosis
* Less than CCyR at 18 months after diagnosis
* Prior accelerated phase or blast phase CML
* Previously documented T315I mutation
* Previous treatment for CML with any other tyrosine kinase inhibitor except for imatinib
* Patients who had any other treatment for CML (transplant) except interferon +/- ara- C, imatinib, hydroxyurea and/or anagrelide
* Impaired cardiac function
* Patients receiving therapy with strong inhibitors of CYP3A4 or medications that prolong the QT interval and cannot be either discontinued or switched to a different medication prior to starting study drug.
* Any other malignancy that is clinically significant or requires active intervention.
* Major surgery within 4 weeks prior to Day 1 of study or who have not recovered from prior surgery
* Treatment with other investigational agents within 30 days of Day 1
* Women who are pregnant, breast feeding, or of childbearing potential without a negative serum test at baseline. Post-menopausal women must be amenorrhoeic for at least 12 months to be considered of non-childbearing potential. Women of childbearing potential must have a negative serum pregnancy test within 7 days of the first dose of nilotinib
* Sexually active male and female patients taking nilotinib unwilling to use adequate contraception throughout the trial and 3 months following discontinuation of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-10-21 (Actual); Primary Completion 2011-05-12 (Actual); Study Completion 2011-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - Comprehensive Cancer Centers of Nevada CCC of Nevada (1), Las Vegas, Nevada
  - Cancer Center of the High Plains, Amarillo, Texas
  - Baylor Health Care System/Sammons Cancer Center Dept. of Sammons Cancer (2), Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 centers in the United States.
Pre-assignment Details: A total of 3 participants were enrolled in the study, of which 1 discontinued the study due to Adverse Event (AE) and 2 participants discontinued as the study got terminated.
Groups:
- Nilotinib: Participants received nilotinib 300 milligram (mg) twice daily (bid) through the mouth (po), every 12 hours in a continuous 28-day cycle up to 2 years.
Period: Overall Study
Arm/Group | Nilotinib
Started | 3
Completed | 0
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — The participants discontinued the study as the study got terminated | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Nilotinib: Participants received nilotinib 300 mg, BID po, every 12 hours in continuous 28-day cycle up to 2 years.
Arm/Group | Nilotinib
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Failure Events up to 2 Years
Description: Treatment failure events from time of study entry in Complete molecular response-Chronic phase (CML-CP) participants with low imatinib trough concentrations less than 850 nanogram per milliliter (<850 ng/mL) treated with nilotinib as defined in European LeukemiaNet (ELN)-guideline.
Time Frame: up to 2 years
Population: The overall number of participants considered for analysis was "0" due to the premature termination of the study and low enrollment; The efficacy and quality of life assessments were not collected and reported in the study.
Arm/Group | Nilotinib
Number analyzed (Participants) | 0

2. Secondary Outcome: European LeukemiaNet (ELN)-Defined Optimal Responses
Time Frame: up to 2 years
Population: as for outcome 1
Arm/Group | Nilotinib
Number analyzed (Participants) | 0

3. Secondary Outcome: Loss of Complete Cytogenetic Response (CCyR), Major Molecular Response (MMR) and Complete Molecular Response (CMR) on Nilotinib
Description: Complete Cytogenetic Response (CCyR) is defined as 0% of Ph+ metaphases. A patient was counted as CCyR at 12 cycles if the patient met the CCyR criteria at the Cycle 12 Visit.
  Major molecular response is defined as values equal or below 0.1% on the International Scale.
  Complete Molecular Response is defined as a Bcr-Abl (a fusion of gene of Bcr and ABl genes) ratio ≤0.0032% on the International Scale Bcr = breakpoint cluster gene Abl = abelson proto-oncogene.
Time Frame: up to 2 years
Population: as for outcome 1
Arm/Group | Nilotinib
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Complete Cytogenetic Response (CCyR), Major Molecular Response (MMR) and Complete Molecular Response (CMR)Achieved on Nilotinib
Description: Durations of major/complete cytogenetic response is defined as the time from the first documentation of the major/ complete response to the first documentation of the disease progression.
Time Frame: up to 2 years
Population: as for outcome 1
Arm/Group | Nilotinib
Number analyzed (Participants) | 0

5. Secondary Outcome: Event-free Survival (EFS), Progression-free Survival (PFS) and Overall Survival (OS) up to 2 Years
Description: Event-free survival was defined as the time from the date of randomization to the date of first occurrence of any of the following events on study treatment: loss of complete hematological response, confirmed loss of complete cytogenetic response (CCyR), confirmed loss of major molecular response (MMR), death from any cause during treatment, progression to the accelerated phase or blast crisis of chronic myelogenous leukemia (CML) per European Leukemia Network (ELN) criteria, whichever was earliest.
  Progressions free survival is defined as time between Day 1 cycle 1 and time to first documented disease progression or death. Disease progression will be determined as per response criteria.
  Overall survival time is defined as the time from the treatment start to the date of death due to any reason.
Time Frame: up to 2 years
Population: as for outcome 1
Arm/Group | Nilotinib
Number analyzed (Participants) | 0

6. Secondary Outcome: European LeukemiaNet (ELN)-Defined Suboptimal Events
Time Frame: up to 2 years
Population: as for outcome 1
Arm/Group | Nilotinib
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants Reported Adverse Events
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Time Frame: up to 2 years
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical examination or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Nilotinib
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=3)
Muscle cramps - legs (Musculoskeletal and connective tissue disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Pruritus Genital (Skin and subcutaneous tissue disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Sore Throat (Infections and infestations) | 1
Mild sweats (General disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes